CLINICAL TRIAL: NCT07330960
Title: Augmenting Existing Normative Data for QbMobile in Healthy Children Aged 6-11 Years.
Status: Not yet recruiting | Type: Observational
Sponsor: Qbtech AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 00091260 QB25-02
Record Dates: First submitted 2025-12-11; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers
  Interventions: Device: Digital software application for cognitive performance and activity measurement (QbMobile, investigational device)

INTERVENTIONS:
Device: Digital software application for cognitive performance and activity measurement (QbMobile, investigational device) — Participants will complete a non-invasive, 10-minute digital tests using the QbMobile Investigational Device. The test objectively measure cognitive performance and activity levels.

SUMMARY:
The purpose of this study is to strengthen the normative QbMobile data for children and adolescents age 6-11 years to allow for a more robust and accurate representation when comparing a patient's QbMobile performance with the appropriate normative reference group.

DETAILED DESCRIPTION:
Participants will be recruited and referred from selected clinics' general population databases, local schools, youth centers and organizations, as well as other general practitioners within the surrounding area.

Participants will be pre-screened via an online questionnaire completed by their parent/legal guardian designed to capture diagnostic history and general demographic information. Access to the questionnaire will be initiated by scanning a QR code on the study flyer that will be visibly posted at locations listed above.

Parents or legal guardians will be asked to provide a reliable phone number within the pre-screening questionnaire, which will be used by the research team to follow up and verify the information submitted in the questionnaire. Once eligibility is confirmed through both the questionnaire and phone verification, participants will be scheduled for enrollment in the study.

On the scheduled study day, participants will complete a 10-minute QbMobile test.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent from parent/legal guardians and assent for all study participants for the QbMobile study;
* Aged > 6 years and < 11 years old;
* Have no documented or suspected current or lifetime diagnosis of ADHD;
* Have adequate sensory and physical ability to complete QbMobile;

Exclusion Criteria:

* Intellectual disability designated by IQ<75;
* Has a concurrent medical diagnosis that could significantly affect test performance such as brain injuries, Parkinson's disease, current epilepsy or active seizures, amyotrophic lateral sclerosis (ALS), multiple sclerosis, dementias (e.g. vascular dementia, Alzheimer disease), unmanaged psychiatric illness;
* Has other conditions that could affect test performance (migraine or other types of severe headache, chronic or acute pain);
* Substance use (e.g., alcohol, drugs) that may affect performance on the day of the tests.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consists of a community-based sample of healthy children aged 6 to 11 years with no history of ADHD. Participants are primarily identified through local schools, community youth organizations, and general practitioners, with additional participants identified through the general patient databases of participating clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Establishment of Normative Statistics for QbMobile Performance | 1 QbMobile test at the clinic visit (Day 1)
  Normative data will be analyzed to generate Standard Deviation (SD) scores and Total Scores for four domains: activity, impulsivity, inattention, and movement patterns. QbMobile SD-scores are standardized metrics derived from the main parameters (attention, impulsivity, activity and movement). These scores are calculated using and age and sex at birth adjusted normative dataset. The QbMobile also produces a Total Score number ranging from 0 to 100, where 0 indicates a low likelihood of exhibiting ADHD symptoms and 100 indicates a high likelihood of exhibiting ADHD symptoms. These scores will enable individual test performance to be expressed relative to normative benchmarks.

SECONDARY OUTCOMES:
Exploratory Analysis of Additional Domain Parameters | 1 QbMobile test at the clinic visit (Day 1)
  Exploratory analyses will be conducted on raw QbMobile data collected at Day 1 to identify potential additional parameters that may serve as indices of activity, attention, impulsivity, and movement from the QbMobile Standard Deviation (SD) Scores and Total Scores. QbMobile SD-scores are standardized metrics derived from the main parameters (attention, impulsivity, activity and movement). These scores are calculated using and age and sex at birth adjusted normative dataset. The QbMobile also produces a Total Score number ranging from 0 to 100, where 0 indicates a low likelihood of exhibiting ADHD symptoms and 100 indicates a high likelihood of exhibiting ADHD symptoms. These parameters will be evaluated for their potential association with ADHD symptomatology.

IPD SHARING:
Plan to Share IPD: No
Due to the nature of the research, limited access to supporting data may be granted upon reasonable request under confidentiality agreements from the corresponding sponsor.